CLINICAL TRIAL: NCT02402309
Title: Phase II Study of the Safety, Pharmacokinetics, and Exploratory Activity of Once Daily (QD) Topical Application of NS2 Cream to Treat Ichthyosis in Subjects With Sjögren-Larsson Syndrome (SLS)
Brief Title: A Study of Topical NS2 Cream to Treat Ichthyosis in Sjögren-Larsson Syndrome (SLS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-003
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Sjögren-Larsson Syndrome
Keywords: Sjögren-Larsson Syndrome; SLS; FALDH Deficiency; Neuro-ichthyosis; Fatty Alcohol:NAD+ Oxidoreductase Deficiency; Fatty Aldehyde Dehydrogenase Deficiency Disease; Congenital Icthyosis Mental Retardation Spasticity Syndrome; Spastic Neurologic Disorder; Oligophrenia; Ichthyosis
MeSH Terms: conditions — Sjogren-Larsson Syndrome; Ichthyosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active topical NS2 1% dermatologic cream (Experimental): NS2 1% topical cream for dermal application
  Interventions: Drug: Active topical NS2 1% dermatologic cream
- Topical vehicle dermatologic (Placebo Comparator): Vehicle placebo for dermal application
  Interventions: Drug: Vehicle placebo 0.0% NS2 dermatologic cream

INTERVENTIONS:
Drug: Active topical NS2 1% dermatologic cream
  Arms: Active topical NS2 1% dermatologic cream
Drug: Vehicle placebo 0.0% NS2 dermatologic cream
  Arms: Topical vehicle dermatologic

SUMMARY:
This is a multi-center, randomized, double-blind, vehicle-controlled, parallel-group study designed to evaluate the safety, pharmacokinetic (PK), and exploratory activity of topically-applied NS2 dermatologic cream administered once-daily (QD) to subjects with ichthyosis secondary to Sjögren- Larsson Syndrome (SLS).

NS2 is expected to trap fatty aldehydes that are pathogenic in SLS patients, and thereby diminish the lipid-aldehyde adduct formation that likely results in ichthyosis associated with SLS, and potentially reduce the mild dermal inflammation characteristic of SLS.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-confirmed diagnosis of SLS
* Active ichthyosis on the lower extremities that is determined to be at least moderate severity

Exclusion Criteria:

* Evidence of an active infection
* Currently receiving immunosuppressive therapy, including intermittent or low-dose corticosteroids and is not able or willing to suspend from 2 weeks before and during the study
* Currently receiving systemic or topical retinoids, other topically applied drugs, or other supplements that could interfere with dermatologic examination findings
* Received an investigational systemic or topically administered drug within 30 days before screening

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B. Rizzo, MD, Principal Investigator — University of Nebraska
Locations (3):
- United States (3):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Penn State Hershey Medical Center - Department of Dermatology, Hershey, Pennsylvania
  - Pediatric and General Dermatology, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical NS2 1% Dermatologic Cream: NS2 1% topical cream for dermal application
  Active topical NS2 1% dermatologic cream
- Topical Vehicle Dermatologic: Vehicle placebo for dermal application
  Vehicle placebo 0.0% NS2 dermatologic cream
Period: Overall Study
Arm/Group | Topical NS2 1% Dermatologic Cream | Topical Vehicle Dermatologic
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical NS2 1% Dermatologic Cream | Topical Vehicle Dermatologic | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.2 (5.08) | 17.3 (5.01) | 15.8 (5.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  White | 3 | 5 | 8
  Other | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Height [Mean (Standard Deviation); unit: centimeters] | 150.0 (19.71) | 157.2 (9.14) | 153.6 (15.13)
Weight [Mean (Standard Deviation); unit: kilograms] | 41.4 (13.07) | 59.8 (14.36) | 50.6 (16.24)
Body Surface Area [Mean (Standard Deviation); unit: Mosteller Method (m2)] | 1.54 (0.527) | 1.95 (0.890) | 1.77 (0.743)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Serious Adverse Event (SAE).
Time Frame: The safety assessment period is approximately 9 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical NS2 1% Dermatologic Cream | Topical Vehicle Dermatologic
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Primary Outcome: Number of Participants Experiencing an Adverse Event Leading to Discontinuation.
Time Frame: The safety assessment period is approximately 9 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical NS2 1% Dermatologic Cream | Topical Vehicle Dermatologic
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was captured for approximately 9 weeks for each subject during clinical trial participation.
Arm/Group | Topical NS2 1% Dermatologic Cream | Topical Vehicle Dermatologic
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topical NS2 1% Dermatologic Cream (N=6) | Topical Vehicle Dermatologic (N=6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes